CLINICAL TRIAL: NCT07122024
Title: Efficacy and Safety of Keverprazan-amoxicillin Dual Therapy for Helicobacter Pylori First-line Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Ye Jun, Professor of Treatment, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Keverprazan Helicobacter pylo; FK2024-6926 (Other Grant/Funding Number: Fosun Pharma)
Record Dates: First submitted 2025-06-03; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Pylori
MeSH Terms: interventions — Amoxicillin; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Keverprazan Dual Therapy for 10 Days (Experimental): Keverprazan 20 mg per dose, twice daily (bid) + Amoxicillin 1 g per dose, three times (tid) daily, for 10 days.
  Interventions: Drug: Keverprazan 10 days
- Keverprazan Dual Therapy for 14 Days (Active Comparator): Keverprazan 20 mg, bid + Amoxicillin 1 g, tid, for 14 days.
  Interventions: Drug: Keverprazan 14 days
- Rabeprazole Quadruple Therapy for 14 Days (Active Comparator): Rabeprazole sodium 10 mg + Amoxicillin 1 g + Clarithromycin 500 mg + Colloidal pectin bismuth 200 mg, bid, for 14 days.
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: Keverprazan 10 days — Keverprazan dual therapy for 10 days (K10 group):
  Keverprazan 20 mg per dose, twice daily (bid) + Amoxicillin 1 g per dose, three times (tid) daily, for 10 days.
  Other Names: Amoxicillin
  Arms: Keverprazan Dual Therapy for 10 Days
Drug: Keverprazan 14 days — Keverprazan dual therapy for 14 days (K14 group): Keverprazan 20 mg, bid + Amoxicillin 1 g, tid, for 14 days.
  Other Names: Amoxicillin
  Arms: Keverprazan Dual Therapy for 14 Days
Drug: Rabeprazole — Rabeprazole quadruple therapy for 14 days (R14 group): Rabeprazole sodium 10 mg + Amoxicillin 1 g + Clarithromycin 500 mg + Colloidal pectin bismuth 200 mg, bid, for 14 days.
  Other Names: Amoxicillin Clarithromycin Colloidal pectin bismuth
  Arms: Rabeprazole Quadruple Therapy for 14 Days

SUMMARY:
This is an open-label, randomized controlled study. The study plans to enroll 414 subjects with Helicobacter pylori infection, who will be randomly assigned to the experimental group (Keverprazan dual therapy for 10 days or Keverprazan dual therapy for 14 days) or the control group (Rabeprazole quadruple therapy for 14 days) at a ratio of 1:1:1.

DETAILED DESCRIPTION:
This is an open-label, randomized controlled study. The study plans to enroll 414 subjects with Helicobacter pylori infection, who will be randomly assigned to the experimental group (Keverprazan dual therapy for 10 days or Keverprazan dual therapy for 14 days) or the control group (Rabeprazole quadruple therapy for 14 days) at a ratio of 1:1:1. Study duration: Starting from the date of ethics approval and clinical registration completion, the project will last for 1 year. If you agree to participate in this study, you will be assigned to one of the three treatment groups through randomization (with a 33% probability for each group), with 138 subjects in each group.

The study is divided into a screening phase and a treatment phase, with a total of 4 visit points:

Screening period: -7 to 0 days

1. Obtain informed consent;
2. Collect demographic information and baseline characteristics of the subject;
3. Record medical history and current treatment, concomitant medications (including prescription and over-the-counter drugs);
4. Vital signs, physical examination;
5. H. pylori test;
6. Review inclusion and exclusion criteria;
7. Eligible subjects will be randomized to receive assigned treatment based on randomization numbers.

Visit period V2 (telephone visit):

K10 group: 10 days (±3 days), K14 group: 14 days (±3 days), R14 group: 14 days (±3 days)

1. Vital signs, physical examination;
2. Record concomitant medications;
3. Record adverse events after medication. Visit period V3: 9 weeks (±7 days)

1) Vital signs, physical examination; 2) H. pylori test; 3) Record concomitant medications; 4) Record adverse events after medication.

ELIGIBILITY:
Inclusion Criteria

1. Adult patients aged 18 to 65 years old, regardless of gender;
2. H. pylori positive, diagnosed a 13C-urea breath test (13C-UBT), ¹⁴C-urea breath test (¹⁴C-UBT), H&E staining or bacterial culture;
3. No previous history of H. pylori eradication therapy;
4. Subjects able to independently complete the recording of the subject diary card;
5. Subjects who fully understand the trial content, voluntarily participate in the trial, can complete the trial process, and sign the informed consent form.

Exclusion Criteria

1. Use of acid-suppressing drugs such as proton pump inhibitors (PPIs), potassium-competitive acid blocker (P-CAB), H2 receptor antagonists, etc., within 2 weeks before enrollment, or use of antibiotics within 4 weeks before enrollment;
2. Active peptic ulcer with complications such as bleeding, perforation, obstruction, canceration, etc.;
3. Previous history of esophageal or gastric surgery;
4. Severe systemic diseases, including diseases of major organs dysfunction such as (cardiac, pulmonary, cerebral), hepatic or renal impairment, malignant neoplasms , or other diseases;
5. Participants with allergies or hypersensitivity to keverprazan, rabeprazole, amoxicillin, clarithromycin, bismuth agents, including its excipients (such as mannitol, microcrystalline cellulose, crospovidone, hypromellose, magnesium stearate, etc.);
6. Female participants who are pregnant, breastfeeding;
7. Long-term alcohol abuse or any other conditions that increase the risk of treatment-related adverse events;
8. Participation in other studies within the past 3 months, inability to clearly express oneself, or inability to cooperate with investigators;
9. Deemed unsuitable for participation in the study by the investigator for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate 6-8 weeks after the end of eradication treatment | 8-10weeks
  Efficacy Endpoints:
  The primary efficacy endpoint is the proportion of subjects achieving successful Helicobacter pylori eradication 6-8 weeks after completion of first-line therapy. Eradication rates will be reported with two-sided 95% confidence intervals (CIs) calculated using the Clopper-Pearson method. Inter-group differences will be estimated along with their 95% CIs using the Miettinen-Nurminen method. Inter-group comparisons will be performed using the chi-square test or Fisher's exact test, as appropriate.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug until 8 weeks after last dose
  Through the incidence, severity (per CTCAE v5.0), and drug-drug interactions of adverse events (AEs) occurring from the start of medication until 8 weeks after the end of medication.

CONTACTS AND LOCATIONS:
Overall Officials: QIN DU, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; JUN YE, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Protocol Inclusion/Exclusion Criteria andFinalStudv Results
Supporting Information: CSR
Time Frame: 2025.12
Access Criteria: Authorization from the PrincipalInvestigator (Pl) of this study is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT07122024/Prot_SAP_000.pdf